CLINICAL TRIAL: NCT01281124
Title: Pilot Phase II Study of 5-Azacytidine in Previously Treated Patients With Advanced NSCLC
Brief Title: Azacitidine in Treating Patients With Previously Treated Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02570; NCI-2011-02570 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000692184; OSU-10100; OSU 10100 (Other: Ohio State University Comprehensive Cancer Center); 8617 (Other: CTEP); N01CM00070 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine

ARMS (1):
- Treatment (azacitidine) (Experimental): Patients receive azacitidine subcutaneously on days 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Diagnostic Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Azacitidine — Given subcutaneously
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II clinical trial is studying how well azacitidine works in treating patients with previously treated advanced non-small cell lung cancer. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the ability of 5-azacytidine to cause DNA hypomethylation and re-expression of silenced tumor suppressor genes when stratified for high or low expression of mir29a, b, and c.

SECONDARY OBJECTIVES:

I. To compare the molecular studies (mir29 expression and tumor suppressor gene methylation) between archival tissue, fresh biopsy pre-treatment samples, and post-treatment fresh samples.

II. To determine the overall response rate by CT (RECIST 1.1 criteria) and PET (EORTC PET response criteria), PFS, and OS of patients treated with azacytidine in the second- or third-line setting.

III. To correlate the blood microRNA profiles (and changes in microRNA profiles) with response to azacytidine.

OUTLINE:

Patients receive azacitidine subcutaneously on days 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tissue and blood sample collection at baseline and periodically during study treatment for correlative studies. After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (stage 4 or recurrent) NSCLC, not eligible for any curative intent treatment

  * Tumor must be histologically or cytologically confirmed
* Measurable disease (as defined by RECIST criteria)
* Patients may have up to two (and at least one) prior cytotoxic regimens in the metastatic setting

  * Prior adjuvant chemotherapy following resection or definitive chemo-radiation for patients with locally advanced disease is not included in this
  * Allowable systemic therapy in the metastatic setting includes 2 cytotoxic regimens and erlotinib and/or other non-cytotoxic drugs (i.e., erlotinib, sorafenib, and other tyrosine kinase inhibitors do not count as a "cytotoxic regimen")
  * Prior adjuvant therapy or definitive chemo-radiation is allowed if completed > six months before the onset of "first-line" therapy in the metastatic setting - in this setting, adjuvant or definitive chemo-radiation will not "count" as one of the two cytotoxic regimens; if however, the patient relapses within six months from completion of adjuvant or definitive chemoradiation, then this therapy will be considered the first-line cytotoxic therapy
  * In the unusual circumstance where patients receive "adjuvant" therapy following resection of oligo-metastatic disease (for example brain metastasis and lung primary resections) and the treating physician decides to administer chemotherapy following all surgery, this will be considered "adjuvant" therapy and the same rules as noted above will apply for initiation of first-line systemic therapy
* No patients with uncontrolled brain metastases or leptomeningeal disease

  * Patients with controlled brain metastases are allowed
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets ≥ 100,000 x 10^9/L
* Hemoglobin ≥ 9.0 gm/100 mL
* Total bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 x ULN
* Creatinine ≤ 1.5 mg/dL OR calculated creatinine clearance > 50 mL/min
* No patients who are pregnant
* Women of childbearing potential must have a negative pregnancy test
* The patient must be willing to use adequate contraception for the duration of study treatment and up to four weeks following the last dose of drug
* Archival diagnostic material sufficient for microRNA evaluation/assessment is preferred, though optional

  * The presence of archival material will not preclude the need for pre and post treatment biopsies
* Willing to undergo biopsy pre-treatment and following first cycle

  * Biopsy may be from any accessible site (primary or metastatic)
* No known HIV or hepatitis B or C (though testing for this is not required)
* No uncontrolled intercurrent illness including, but not limited to:

  * Symptomatic CHF
  * Unstable angina pectoris
  * Serious cardiac arrhythmia
  * Serious infection
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No patients who have significant psychiatric illness that, in the opinion of the principal investigator, would prevent adequate informed consent or render therapy unsafe
* Patients may not have had a prior invasive malignancy except for adequately treated non-melanoma cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 2 years

  * For example, a stage 1 (T1c) prostate cancer 2 years prior to a diagnosis of NSCLC would not be exclusionary, however, a metastatic prostate cancer currently receiving hormonal or chemotherapy would be excluded
* No other concurrent palliative radiotherapy
* Recovered from prior surgery, radiation, or chemotherapy to ≤ grade 2 toxicity
* Palliative radiation or surgical procedures (for example, endobronchial therapy) is allowed, but must have been completed > 2 weeks prior to starting treatment
* No other investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01-12 (Actual); Primary Completion 2011-04-15 (Actual); Study Completion 2012-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Otterson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (5-Azacytidine): Patients receive 5-azacitidine subcutaneously at the starting dose level of 75 mg/m2 on an outpatient basis daily for 7 days on a 28 day cycle.
Period: Overall Study
Arm/Group | Treatment (5-Azacytidine)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Azacitidine)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: DNA Hypomethylation and Re-expression of Silenced Tumor Suppressor Genes When Stratified for Low or High Expression of mir29
Description: The change in mean methylation of the genes between the patients with a low mir29 and a high mir29 expression will be evaluated by a two-sample t-test. Secondary analyses include a multivariate regression where all 5 changes in methylation will be regressed on mir29 expression (low vs. high) and adjusted for patient demographic and clinical attributes at baseline.
Time Frame: Up to 12 weeks after completion of study treatment
Population: Data analysis was not done due to low accrual for this trial.
Groups:
- Treatment (5-Azacyitidine): Patients receive azacitidine subcutaneously on days 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (5-Azacyitidine)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Analyzed using a Kaplan-Meier methods.
Time Frame: From the day of initial treatment until death (from any cause), assessed up to 12 weeks after completion of study treatment
Population: Data analysis was not done due to low accrual for this trial.
Groups:
- Treatment (5-Azacytidine): Patients receive azacitidine subcutaneously on days 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (5-Azacytidine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: Analyzed using a Kaplan-Meier methods.
Time Frame: From the day of initial treatment until documented disease progression (per PET) or death, assessed up to 12 weeks after completion of study treatment
Population: Data analysis was not done due to low accrual for this trial.
Arm/Group | Treatment (Azacitidine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline through end of follow up period (12 weeks after removal from study or until death, whichever occurs first).
Description: Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.
Arm/Group | Treatment (Azacitidine)
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine) (N=1)
Cardiac Arrest (Cardiac disorders) | 1 (1) — event occurred after removal from study
Pericardial effusion (Cardiac disorders) | 1 (1) — event occured after removal from study
Pericardial tamponade (Cardiac disorders) | 1 (1) — event occured after removal from study
Lymphocyte count decreased (Investigations) | 1 (1) — event occured after removal from study
Anorexia (Metabolism and nutrition disorders) | 1 (1) — event occured after removal from study
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) — event occured after removal from study
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) — event occured after removal from study
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — event occured after removal from study
Insomnia (Psychiatric disorders) | 1 (1) — event occured after removal from study
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — event occured after removal from study
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — event occured after removal from study
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine) (N=1)
Urticaria (Welts) (Skin and subcutaneous tissue disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia-Viral (Infections and infestations) | 1 (1)
Lymphopenia (Investigations) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to low enrollment of this trial all outcomes were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less